CLINICAL TRIAL: NCT04392726
Title: Ultra-Low Dose Computed Tomography For Diagnosis And Follow-Up Of Patients With Diffuse Parenchymal Lung Disease (DPLD)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Liran Levy, Transplant pulmonologist, Sheba Medical Center
Other Study IDs: SHEBA-20-7020-20-SMC-LL-CTIL
Record Dates: First submitted 2020-03-22; First posted 2020-05-19 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Diffuse Parenchymal Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with suspected DPLD
- patients with known DPLD

SUMMARY:
The primary intention of this study is to determine the diagnostic performance of ultra-low-dose CT (ULDCT) in diagnosis and follow-up of diffuse parenchymal lung disease (DPLD). We hypothesize that inspiratory and expiratory chest ULDCT has comparable diagnostic yield to standard dose chest High-resolution computed tomography (HRCT) and utility for follow-up of patients with known DPLD. We will study this hypothesis through the following aims:

1. Determine whether inspiratory and expiratory ULDCT are comparable to HRCT in identifying mosaic attenuation due to air-trapping.
2. Determine whether ULDCT is as good as HRCT for follow-up of patients with established DPLD to identify disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. suspected or known DPLD
2. referred to DPLD observation

Exclusion Criteria:

1. other lung related diseases

-

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with known or suspected DPLD
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure of this study is to determine the diagnostic performance of ULDCT in diagnosis of DPLD. | during the procedure/surgery
  The diagnostic performance will be evaluated according to the biopsy results
The primary outcome measure of this study is to determine the prognostic performance of ULDCT in the follow up of DPLD. | during the procedure/surgery
  The diagnostic performance will be evaluated according to the biopsy results

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel